CLINICAL TRIAL: NCT03943823
Title: Postmenopausal Pessary Users: Estrogen Versus Trimosan
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulties in recruiting and retaining patients due to the COVID pandemic; lack of availability of study drug trimosan; lack of study personnel
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Gazala Siddiqui, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-15-0337
Record Dates: First submitted 2019-05-07; First posted 2019-05-09 (Actual); Results first posted 2023-03-01 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Vaginosis; Vaginosis, Bacterial; Vaginal Discharge
Keywords: Pessary; Vaginal pH
MeSH Terms: conditions — Vaginal Diseases; Vaginosis, Bacterial; Vaginal Discharge

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Estrogen vaginal cream (Active Comparator)
  Interventions: Drug: Estrogen vaginal cream
- Trimo-San vaginal gel (Active Comparator)
  Interventions: Drug: Trimo-San vaginal gel

INTERVENTIONS:
Drug: Estrogen vaginal cream — Either Premarin or Estrace cream will be used (dependent on patient's insurance). Premarin 1 gram every night for the first 7 days, then 0.5 grams twice weekly. Estrace cream 2 grams daily for first 7 days, then 1 gram twice-weekly.
  Other Names: Estrace Cream; Premarin Cream
  Arms: Estrogen vaginal cream
Drug: Trimo-San vaginal gel — Half applicator for three times a week for 1st week, then half applicator for 2 times a week.
  Other Names: Trimo-San
  Arms: Trimo-San vaginal gel

SUMMARY:
The purpose of the study is to compare vaginally applied estrogen with the vaginal gel trimosan for their effects on vaginal pH and vaginal symptoms in postmenopausal pessary users.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal female pessary user (ring with support pessaries only). Postmenopausal will be defined as: amenorrhea for a year or 3 months after surgical bilateral salpingo-oophorectomy
* Is a new pessary user, or has not had a pessary for a year

Exclusion Criteria:

* Pregnancy
* Persistent Bacterial Vaginosis infection in the first two clinic encounters
* Currently on hormone replacement therapy
* Previously on hormone replacement therapy in the past 6 months
* Currently on antibiotics
* Patients with existing vaginal erosions/ulcerations

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-05-07 (Actual); Primary Completion 2021-03-08 (Actual); Study Completion 2021-04-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gazala Siddiqui, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Estrogen Vaginal Cream | Trimo-San Vaginal Gel
Started | 2 | 2
Completed | 1 | 2
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Estrogen Vaginal Cream | Trimo-San Vaginal Gel | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Customized [Count of Participants; unit: Participants]
  age 60 to 75 | 2 | 2 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 0 | 1 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Vaginal pH as Measured by pH Strips
Description: pH is measured on a scale of 0 to 14, with lower values indicating greater acidity and higher values indicating greater alkalinity.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Estrogen Vaginal Cream | Trimo-San Vaginal Gel
Number analyzed (Participants) | 2 | 2
pH | 4.5 (0.70) | 6 (0)

2. Primary Outcome: Vaginal pH as Measured by pH Strips
Description: as for outcome 1
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Estrogen Vaginal Cream | Trimo-San Vaginal Gel
Number analyzed (Participants) | 2 | 2
pH | 4.25 (.35) | 5 (.70)

3. Secondary Outcome: Number of Participants Who Exhibited Vaginal Symptoms as Assessed by a Questionnaire
Time Frame: baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Estrogen Vaginal Cream | Trimo-San Vaginal Gel
Number analyzed (Participants) | 2 | 2
Participants | 1 | 0

4. Secondary Outcome: Number of Participants Who Exhibited Vaginal Symptoms as Assessed by a Questionnaire
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Estrogen Vaginal Cream | Trimo-San Vaginal Gel
Number analyzed (Participants) | 2 | 2
Participants | 1 | 0

5. Other Pre Specified Outcome: Number of Participants With Vaginitis Infection
Description: Presence of vaginitis infection will be assessed with an Affirm test, which probes for Gardnerella vaginalis, Candida albicans, and Trichomonas vaginalis.
Time Frame: baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Estrogen Vaginal Cream | Trimo-San Vaginal Gel
Number analyzed (Participants) | 2 | 2
Participants
  Gardnerella vaginalis | 1 | 2
  Candida albicans | 2 | 0
  Trichomonas vaginalis | 0 | 0

6. Other Pre Specified Outcome: Number of Participants With Vaginitis Infection
Description: as for outcome 5
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Estrogen Vaginal Cream | Trimo-San Vaginal Gel
Number analyzed (Participants) | 2 | 2
Participants
  Gardnerella vaginalis | 2 | 2
  Candida albicans | 2 | 0
  Trichomonas vaginalis | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Estrogen Vaginal Cream | Trimo-San Vaginal Gel
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2

LIMITATIONS AND CAVEATS:
Early termination as a result of discontinuation of in-person research due to COVID-19 pandemic, as well as unavailability of study drug.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-09-28): https://cdn.clinicaltrials.gov/large-docs/23/NCT03943823/Prot_SAP_000.pdf